CLINICAL TRIAL: NCT00269230
Title: Attain StarFix™ Model 4195 Left Ventricular Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: CRDM Core Clinical, Medtronic CRDM
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 234
Expanded Access: Available
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-10

CONDITIONS: Heart Failure
Keywords: cardiac resynchronization therapy, left ventricular Lead, Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pacing Lead — Left ventricular pacing lead

SUMMARY:
People who have abnormal heart beats, or whose heart does not beat on its own, may need an electronic device called a pacemaker or a defibrillator. Furthermore, people whose hearts have a reduced pumping ability may need a device are called cardiac resynchronization therapy (CRT) device. A CRT device is implanted surgically just under the skin in the upper chest area. This device then helps the heart beat at a regular rhythm by sending electrical signals (pacing) directly to the heart tissue through flexible wires called leads. The device may also be able to stop the heart from beating too fast. Three leads are implanted into the chambers of your heart. Two of the leads will be placed on the right side of your heart. The third lead is placed on the left side of your heart and is the lead being studied.

The purpose of this study is to evaluate the safety and efficacy of the Attain StarFixTM Model 4195 Left Ventricular (LV) Lead. This particular model lead has special characteristics that may help to better keep it in position once it is implanted into the left ventricle. It is also "steroid-eluting" which means that over time it slowly releases a small amount of medication into the heart tissue to help prevent too much swelling around the area it is implanted.

ELIGIBILITY:
Inclusion Criteria:

* QRS > 130 ms (The QRS interval is a measurement of how the electrical signal involved in a heart beat travels, or is conducted, through the ventricles. A wide QRS (more than 120) suggests that there is a conduction problem, or block, in the ventricles.)
* Left Ventricular Ejection Fraction (EF) < 35% (Ejection Fraction is a measurement of how well the left ventricle pumps blood out to the rest of the body. The higher the EF the more blood the ventricle is pumping.)
* Subject has moderate to severe heart failure despite medications

Exclusion Criteria:

* Subjects with a previous lead in the left ventricle or previous implant attempt within 30 days of implant or ongoing complications from a previous unsuccessful attempt
* Subjects with chest pain or who have had a heart attack within the past month before enrollment in the study
* Subjects that have had certain surgeries on their heart within the past three months
* Subjects with chronic (permanent) fast heart beats in the upper chambers of the heart (atrial arrhythmias)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2004-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy at 3 months | 3 Months

SECONDARY OUTCOMES:
Implant success rate and times with the Model 4195; Handling characteristics and electrical performance of the Model 4195; All adverse events occurring throughout study | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Stuart W Adler II, MD, Principal Investigator — St. Paul Heart Clinic
Locations (25):
- United States (20):
  - Long Beach, California
  - Palo Alto, California
  - Newark, Delaware
  - Jacksonville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Lexington, Kentucky
  - Grand Rapids, Michigan
  - Saginaw, Michigan
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Newark, New Jersey
  - Rochester, New York
  - Durham, North Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Temple, Texas
  - Milwaukee, Wisconsin
- Canada (4):
  - Calgary, Alberta
  - Victoria, British Columbia
  - London, Ontario
  - Sainte-Foy, Quebec
- Milan, Italy